CLINICAL TRIAL: NCT02579590
Title: Evaluation of Female Sexual Functions in Progestogen-only Contraceptive Users
Brief Title: The Female Sexual Functions With Progestogen-only Contraception
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Other Study IDs: AFSFI
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Female Sexual Function
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DEMPA group: This group are using DMPA (Depot Medroxyprogesterone Acetate 150 mg) injection every 3 month for 6-12 month
  Interventions: Drug: Depot Medroxyprogesterone Acetate 150 mg
- Implanon group: This group are using "Implanon " (etonogestrel implant) 68 mg implant for 6-12 month
  Interventions: Drug: Implanon( 68 mg etonogestrel implant)
- Cerazette group: This group are using Cerazette pills (75 micrograms desogestrel) one pill every day for 28 days without pill-free interval for 6-12 month.
  Interventions: Drug: Cerazette pills (75 micrograms desogestrel)
- Normal healthy group: Those women not using any method of contraception

INTERVENTIONS:
Drug: Depot Medroxyprogesterone Acetate 150 mg — the DMPA user" where they are using Depot Medroxyprogesterone Acetate 150 mg (DMPA; Phrmcia) injection every 3 month
  Groups: DEMPA group
Drug: Implanon( 68 mg etonogestrel implant) — where they are using etonogestrel 68 mg implant (Implanon; Organon)
  Groups: Implanon group
Drug: Cerazette pills (75 micrograms desogestrel) — where they are using desogestrel 75 micrograms (Cerazette; Organon), one pill every day for 28 days without pill-free interval.
  Groups: Cerazette group

SUMMARY:
Female sexual dysfunction is age-related, progressive, and very common condition. The physiology of the female sexual function is a complex condition affected by emotional, medical and hormonal elements.

Progestogen-only contraception relies on progestogens alone to achieve contraception. There are several progestogen only contraceptive methods include progestogen only pill (minipill), subdermal implants, Depo-Provera (DMPA) and levonorgestrel intrauterine system. Many studies in literature reported the negative effect of combined oral contraceptive pills (COCs) on female sexual function due to decrease in bioavailability of testosterone and increase level of sex hormone binding globulin (SHBG) which leads to decrease in free testosterone level contributes to dysfunction.

However, the progesterone only methods contains no estrogen, so it has less effect on sex hormone binding globulin and therefore less effect on free testosterone. DMPA (injectable progestins) is an injectable progestin is a highly reliable form of contraception. Nelson in 1996 found that about 6% of women using DMPA reported either lost or decreased libido. More recent study by Fortenberry in 2011 reported that DMPA had no effect on sexual interest compared with nonusers of any hormonal method of contraception in an adolescent population. The etonogestrel implant (Implanon) is a single rod that is inserted into the medial side of non dominant upper arm. Although in general, it is very effective and has relatively low side effect, a decreased libido has been noted.

Cerazette is a progestogen-only contraceptive pill containing 75 micrograms of desogestrel. It acts mainly by inhibiting ovulation. Cerazette users also may complain of decreased libido.

The estrogen is the main hormone which responsible for vitality of the pelvic organ especially the vagina. The main mechanism of action of the DMPA, Implanon and Cerazette is inhibition of ovulation, which leads to decrease in the estrogen level, which causes a drop in blood flow in uterine artery and accordingly the vagina artery. That can affect vaginal lubrication, causing the vagina to be too dry for comfortable sex.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 20-45 years old.
* Sexually active women with regular marital life.
* Using DMPA, Implanon or Cerazette for at least 6 months and no more than 12 months.
* Using the above method only for pregnancy prevention.
* Have not any medical or gynaecologic problem.

Exclusion Criteria:

* Lactating women
* Women have abnormal uterine bleeding with contraception

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants will be recruited from the Outpatient Family planning Clinic of the Women's Health Hospital in the period between the first of November 2015 and the first of May 2016. All recruited women are using injectable progestin (DMPA), subdermal implant (Implanon) or progesterone only pills (Cerazette) for 6-12 months.
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Female Sexual function | 6 months
  The investigators will assess the female sexual function by Arabic Female Sexual Function Index (AFSFI) which is a brief and validated questionnaire designed to assess the sexual functioning in a many Arabic countries during the past month. if the score < 28.1; this will mean female sexual dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Ali, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes